CLINICAL TRIAL: NCT01985763
Title: Genistein Combined With FOLFOX or FOLFOX-Avastin for Treatment of Metastatic Colorectal Cancer: Phase I/II Pilot Study
Brief Title: Genistein in Treatment of Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sofya Pintova (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Sofya Pintova, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-1697
Record Dates: First submitted 2013-11-09; First posted 2013-11-15 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: Colon Cancer; Rectal Cancer; Colorectal Cancer
Keywords: Genistein; soy supplements; phytoestrogens; colon cancer; rectal cancer; colorectal cancer; metastatic; stage IV; FOLFOX; FOLFOX-Avastin; Chemotherapy
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis | interventions — Genistein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Genistein (Experimental): Genistein combined with FOLFOX or FOLFOX-Avastin Genistein 60mg/day orally for 7 days every 2 weeks. Genistein will be administered beginning 4 days prior to FOLFOX or FOLFOX-Avastin and continuing the 3 days of chemotherapy.
  Interventions: Drug: Genistein

INTERVENTIONS:
Drug: Genistein — Genistein combined with FOLFOX or FOLFOX-Avastin
  Other Names: Bonistein

SUMMARY:
Colorectal neoplasms are the third most common malignancies in the United States. Patients with metastatic (stage IV) colorectal cancer have a median life expectancy of 2 years. The response rates to chemotherapy range from 35-40%.

Epidemiologic evidence suggests that soy compounds may reduce the incidence of colorectal cancers. Laboratory analyses demonstrate that genistein, a soy-derived compound, may inhibit Wnt signaling, a pathway activated in majority of colorectal cancers. Laboratory observations also demonstrate that genistein may augment growth inhibition when combined with chemotherapeutic agents of 5-Fluorouracil and platinum compounds.

Based on pre-clinical data the investigators hypothesize that combining genistein with the standard of care chemotherapeutic regimens will reduce chemotherapy resistance and improve response rates in patients. The aim of the study is to add genistein to the regimens of FOLFOX or FOLFOX-Avastin in patients with newly diagnosed stage IV colon or rectal neoplasms.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the tolerability of genistein when combined with chemotherapy

Secondary:

* Evaluate Response Rate (RR) as measured by the radiologic RECIST criteria
* Evaluate Progression Free Survival (PFS)

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients ≥18 years old
* Have pathologically confirmed colon or rectal carcinoma
* Have metastatic (stage IV) disease
* Have a plan by treating physician to receive FOLFOX or FOLFOX-Avastin
* Have an Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Have adequate hematopoietic, hepatic and renal function

  1. Hematopoietic function

     * Hemoglobin ≥10g/dL
     * Absolute Neutrophil Count(ANC) ≥1,500cells/mm2
     * Platelet Count ≥100,000/µL
  2. Hepatic Function

     * Total bilirubin ≤ 1.5x the upper limit of normal
     * ALT and AST must each be ≤2,5x the upper limits of normal
  3. Renal Function

     * Estimated creatinine clearance (Clcr) ≥30 mL/minute
* Are not pregnant and do not plan to become pregnant

Exclusion Criteria:

* Prior systemic chemotherapy for metastatic disease
* History of breast cancer, endometrial cancer or ovarian cancer or taking aromatase inhibitors or selective estrogen receptor modulators
* Patients taking MAO-inhibitors
* History of myocardial infarctions or cardiac stent placement less than 1 year before recruitment into the study
* Unable to give informed consent or comply with clinical trial requirements
* Uncontrolled hypertension
* History of clinically significant GI bleeding within prior 2 months prior to enrollment
* Presence of GI fistula
* Prior history of bowel perforation
* History of CNS thrombotic/embolic or ischemic events
* Have past or current, acute or chronic concurrent medical condition/illness or therapy that, in the opinion of the investigator, would make the subject unsuitable for the clinical trial or unable to comply with the follow up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-11; Primary Completion 2017-01-19 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall F Holcombe, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Sofya Pintova, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] DeCosse JJ, Ngoi SS, Jacobson JS, Cennerazzo WJ. Gender and colorectal cancer. Eur J Cancer Prev. 1993 Mar;2(2):105-15. doi: 10.1097/00008469-199303000-00003. PMID 8461861
- [Background] Hebert-Croteau N. A meta-analysis of hormone replacement therapy and colon cancer in women. Cancer Epidemiol Biomarkers Prev. 1998 Aug;7(8):653-9. PMID 9718216
- [Background] Haenszel W, Berg JW, Segi M, Kurihara M, Locke FB. Large-bowel cancer in Hawaiian Japanese. J Natl Cancer Inst. 1973 Dec;51(6):1765-79. doi: 10.1093/jnci/51.6.1765. No abstract available. PMID 4797262
- [Background] Hu JF, Liu YY, Yu YK, Zhao TZ, Liu SD, Wang QQ. Diet and cancer of the colon and rectum: a case-control study in China. Int J Epidemiol. 1991 Jun;20(2):362-7. doi: 10.1093/ije/20.2.362. PMID 1917235
- [Background] Nishi M, Yoshida K, Hirata K, Miyake H. Eating habits and colorectal cancer. Oncol Rep. 1997 Sep-Oct;4(5):995-8. doi: 10.3892/or.4.5.995. PMID 21590181
- [Background] Kono S, Imanishi K, Shinchi K, Yanai F. Relationship of diet to small and large adenomas of the sigmoid colon. Jpn J Cancer Res. 1993 Jan;84(1):13-9. doi: 10.1111/j.1349-7006.1993.tb02777.x. PMID 8449821
- [Background] Witte JS, Longnecker MP, Bird CL, Lee ER, Frankl HD, Haile RW. Relation of vegetable, fruit, and grain consumption to colorectal adenomatous polyps. Am J Epidemiol. 1996 Dec 1;144(11):1015-25. doi: 10.1093/oxfordjournals.aje.a008872. PMID 8942431
- [Background] Pereira MA, Barnes LH, Rassman VL, Kelloff GV, Steele VE. Use of azoxymethane-induced foci of aberrant crypts in rat colon to identify potential cancer chemopreventive agents. Carcinogenesis. 1994 May;15(5):1049-54. doi: 10.1093/carcin/15.5.1049. PMID 8200067
- [Background] Helms JR and Gallaher DD, The effect of dietary soy protein isolate and genistein on the development of preneoplastic lesions (aberrant crypts) in rats. 1995 Cancer Lett:125
- [Background] Thiagarajan DG, Bennink MR, Bourquin LD, Kavas FA. Prevention of precancerous colonic lesions in rats by soy flakes, soy flour, genistein, and calcium. Am J Clin Nutr. 1998 Dec;68(6 Suppl):1394S-1399S. doi: 10.1093/ajcn/68.6.1394S. PMID 9848506
- [Background] Li Y, Ahmed F, Ali S, Philip PA, Kucuk O, Sarkar FH. Inactivation of nuclear factor kappaB by soy isoflavone genistein contributes to increased apoptosis induced by chemotherapeutic agents in human cancer cells. Cancer Res. 2005 Aug 1;65(15):6934-42. doi: 10.1158/0008-5472.CAN-04-4604. PMID 16061678
- [Background] Linsalata M, Russo F, Notarnicola M, Guerra V, Cavallini A, Clemente C, Messa C. Effects of genistein on the polyamine metabolism and cell growth in DLD-1 human colon cancer cells. Nutr Cancer. 2005;52(1):84-93. doi: 10.1207/s15327914nc5201_11. PMID 16091008
- [Background] Qi W, Weber CR, Wasland K, Savkovic SD. Genistein inhibits proliferation of colon cancer cells by attenuating a negative effect of epidermal growth factor on tumor suppressor FOXO3 activity. BMC Cancer. 2011 Jun 3;11:219. doi: 10.1186/1471-2407-11-219. PMID 21639915
- [Background] Miyaki M, Konishi M, Kikuchi-Yanoshita R, Enomoto M, Igari T, Tanaka K, Muraoka M, Takahashi H, Amada Y, Fukayama M, et al. Characteristics of somatic mutation of the adenomatous polyposis coli gene in colorectal tumors. Cancer Res. 1994 Jun 1;54(11):3011-20. PMID 8187091
- [Background] Zhang Y, Chen H. Genistein attenuates WNT signaling by up-regulating sFRP2 in a human colon cancer cell line. Exp Biol Med (Maywood). 2011 Jun 1;236(6):714-22. doi: 10.1258/ebm.2011.010347. Epub 2011 May 13. PMID 21571909
- [Background] Hwang JT, Ha J, Park OJ. Combination of 5-fluorouracil and genistein induces apoptosis synergistically in chemo-resistant cancer cells through the modulation of AMPK and COX-2 signaling pathways. Biochem Biophys Res Commun. 2005 Jul 1;332(2):433-40. doi: 10.1016/j.bbrc.2005.04.143. PMID 15896711
- [Background] Solomon LA, Ali S, Banerjee S, Munkarah AR, Morris RT, Sarkar FH. Sensitization of ovarian cancer cells to cisplatin by genistein: the role of NF-kappaB. J Ovarian Res. 2008 Nov 24;1(1):9. doi: 10.1186/1757-2215-1-9. PMID 19025644
- [Background] Yanhong H, et al, Genistein sensitizes ovarian carcinoma cells to chemotherapy by switching the cell cycle progression in vitro. J Medical Colleges of PLA:125-135
- [Background] Saltz LB, Clarke S, Diaz-Rubio E, Scheithauer W, Figer A, Wong R, Koski S, Lichinitser M, Yang TS, Rivera F, Couture F, Sirzen F, Cassidy J. Bevacizumab in combination with oxaliplatin-based chemotherapy as first-line therapy in metastatic colorectal cancer: a randomized phase III study. J Clin Oncol. 2008 Apr 20;26(12):2013-9. doi: 10.1200/JCO.2007.14.9930. PMID 18421054
- [Background] Metzner JE, Frank T, Kunz I, Burger D, Riegger C. Study on the pharmacokinetics of synthetic genistein after multiple oral intake in post-menopausal women. Arzneimittelforschung. 2009;59(10):513-20. doi: 10.1055/s-0031-1296435. PMID 19998579
- [Background] Setchell KD, Faughnan MS, Avades T, Zimmer-Nechemias L, Brown NM, Wolfe BE, Brashear WT, Desai P, Oldfield MF, Botting NP, Cassidy A. Comparing the pharmacokinetics of daidzein and genistein with the use of 13C-labeled tracers in premenopausal women. Am J Clin Nutr. 2003 Feb;77(2):411-9. doi: 10.1093/ajcn/77.2.411. PMID 12540402
- [Background] Takimoto CH, Glover K, Huang X, Hayes SA, Gallot L, Quinn M, Jovanovic BD, Shapiro A, Hernandez L, Goetz A, Llorens V, Lieberman R, Crowell JA, Poisson BA, Bergan RC. Phase I pharmacokinetic and pharmacodynamic analysis of unconjugated soy isoflavones administered to individuals with cancer. Cancer Epidemiol Biomarkers Prev. 2003 Nov;12(11 Pt 1):1213-21. PMID 14652284
- [Background] Fischer L, Mahoney C, Jeffcoat AR, Koch MA, Thomas BE, Valentine JL, Stinchcombe T, Boan J, Crowell JA, Zeisel SH. Clinical characteristics and pharmacokinetics of purified soy isoflavones: multiple-dose administration to men with prostate neoplasia. Nutr Cancer. 2004;48(2):160-70. doi: 10.1207/s15327914nc4802_5. PMID 15231450
- [Background] Ullmann U, Oberwittle H, Grossmann M, Riegger C. Repeated oral once daily intake of increasing doses of the novel synthetic genistein product Bonistein in healthy volunteers. Planta Med. 2005 Oct;71(10):891-6. doi: 10.1055/s-2005-864186. PMID 16254818
- [Background] Busby MG, Jeffcoat AR, Bloedon LT, Koch MA, Black T, Dix KJ, Heizer WD, Thomas BF, Hill JM, Crowell JA, Zeisel SH. Clinical characteristics and pharmacokinetics of purified soy isoflavones: single-dose administration to healthy men. Am J Clin Nutr. 2002 Jan;75(1):126-36. doi: 10.1093/ajcn/75.1.126. PMID 11756070
- [Derived] Pintova S, Dharmupari S, Moshier E, Zubizarreta N, Ang C, Holcombe RF. Genistein combined with FOLFOX or FOLFOX-Bevacizumab for the treatment of metastatic colorectal cancer: phase I/II pilot study. Cancer Chemother Pharmacol. 2019 Sep;84(3):591-598. doi: 10.1007/s00280-019-03886-3. Epub 2019 Jun 15. PMID 31203390

RESULTS

PARTICIPANT FLOW:
Groups:
- Genistein: Genistein combined with FOLFOX or FOLFOX-Avastin Genistein 60mg/day orally for 7 days every 2 weeks. Genistein administered beginning 4 days prior to FOLFOX or FOLFOX-Avastin and continuing the 3 days of chemotherapy.
Period: Overall Study
Arm/Group | Genistein
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Genistein
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 61 [32 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 7
ECOG [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) measures level of functioning in terms of daily living abilities:
  0-Fully active, able to carry on all pre-disease performance without restriction
  1-Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg.light house work
  Participants
    0 | 8
    1 | 5
Tumor Location [Count of Participants; unit: Participants]
  Right Colon | 3
  Left Colon | 10
KRAS/NRAS [Count of Participants; unit: Participants]
  Wild Type (WT) | 5
  Mutated | 6
  Unknown | 2
BRAF V600F [Count of Participants; unit: Participants]
  WT | 11
  Mutated | 0
  Unknown | 2
Number of Metastatic Sites [Count of Participants; unit: Participants]
  1 | 8
  2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Number of adverse events to assess tolerability of genistein treatment. Evaluation of side effects conducted every 14 days before each chemotherapy/genistein cycle.
Time Frame: up to 6 months
Measure: Number; unit: events
Arm/Group | Genistein
Number analyzed (Participants) | 13
events
  Grade 1 | 250
  Grade 2 | 119
  Grade 3 | 24
  Grade 4 | 0

2. Primary Outcome: Percent Change in Tumor Size
Description: Percent change in tumor size after cycle 6. Each cycle is 21 days.
Time Frame: end of Cycle 6
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Genistein
Number analyzed (Participants) | 13
Percent change | -43.0 [-49.8 to -1.3]

3. Secondary Outcome: Response Rate RECIST Criteria
Description: Response Rate (RR) as measured by radiologic RECIST criteria. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: end of Cycle 6
Measure: Count of Participants; unit: Participants
Arm/Group | Genistein
Number analyzed (Participants) | 13
Participants
  PR | 8
  SD | 1
  PD | 2
  Not evaluable | 2

4. Secondary Outcome: Number of Participants With an Overall Response Rate (ORR)
Description: Number of participants with an ORR - the portion of patients with a tumor size reduction of a predefined amount for a minimum time period
Time Frame: up to 50 months
Measure: Count of Participants; unit: Participants
Arm/Group | Genistein
Number analyzed (Participants) | 13
Participants | 6

5. Secondary Outcome: Best Overall Response Rate RECIST Criteria
Description: Best Overall Response Rate (ORR) as measured by radiologic RECIST criteria. The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started). In general, the patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.
  SD - target lesion SD, non target lesions Non-PD, and no new lesions. PR - target lesion CR, non target lesions Incomplete response/SD and no new lesions; or target lesion PR, non target lesions Non-PD, and no new lesions.
  PD - target lesions PD, non target lesions Any, can have new lesions; or target lesions Any, non target lesions PD, can have new lesions; or target lesions Any, non target lesions Any, have new lesions.
Time Frame: up to 50 months
Measure: Count of Participants; unit: Participants
Arm/Group | Genistein
Number analyzed (Participants) | 13
Participants
  PR | 6
  SD | 3
  PD | 2
  Not evaluable | 2

6. Secondary Outcome: Number of Participants With Best Overall Response Rate (ORR)
Description: The number of participants with best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started). In general, the patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.
Time Frame: up to 50 months
Measure: Count of Participants; unit: Participants
Arm/Group | Genistein
Number analyzed (Participants) | 13
Participants | 8

7. Secondary Outcome: Progression Free Survival (PFS)
Description: Patients monitored for progression. Progression-free survival (PFS) is the length of time during and after the treatment that a patient lives with the disease but it does not get worse.
Time Frame: up to 50 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Genistein
Number analyzed (Participants) | 13
months | 11.5 [4.9 to 21.7]

8. Secondary Outcome: Percent of Patients With Progression Free Survival (PFS) at 6 Months and 12 Months
Description: Patients monitored for progression during the study period and 1 year following.
  Progression-free survival (PFS) is the length of time during and after the treatment that a patient lives with the disease but it does not get worse.
Time Frame: 6 month and 12 month
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genistein
Number analyzed (Participants) | 13
percentage of participants
  6 months | 69 [48 to 99]
  12 months | 38 [19 to 76]

9. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival - Number of months still living since baseline
Time Frame: up to 50 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Genistein
Number analyzed (Participants) | 13
months | 36.5 [29.5 to 50]

ADVERSE EVENTS:
Time Frame: 6 months
Description: AEs collected for when subjects on Genistein alone and when subjects on Genistein and Chemotherapy
Groups:
- Genistein: Genistein 60mg/day orally for 4 days before chemotherapy.
- Genistein and Chemotherapy: Genistein combined with FOLFOX or FOLFOX-Avastin Genistein 60mg/day orally for 7 days every 2 weeks. Genistein administered beginning 4 days prior to chemotherapy.
Arm/Group | Genistein | Genistein and Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genistein (N=13) | Genistein and Chemotherapy (N=13)
Fatigue (General disorders) | 2 (6) | 11 (55)
Hot Flashes (General disorders) | 2 (8) | 1 (1)
Mucositis (General disorders) | 0 (0) | 5 (11)
Hypertension (Cardiac disorders) | 1 (2) | 12 (88)
Rash (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 6 (23)
Nausea (Gastrointestinal disorders) | 2 (10) | 8 (27)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (9)
Bleeding (Blood and lymphatic system disorders) | 1 (1) | 6 (12)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thromboembolism (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cold Sensitivity (Nervous system disorders) | 0 (0) | 12 (55)
Headache (Nervous system disorders) | 4 (11) | 1 (1)
Neuropathy (Nervous system disorders) | 2 (2) | 7 (34)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 8
Anorexia (Gastrointestinal disorders) | 0 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 8
Constipation (Gastrointestinal disorders) | 1 | 2
Fever (Infections and infestations) | 0 | 1
GERD (Gastrointestinal disorders) | 0 | 8 — Gastroesophageal reflux disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT01985763/Prot_000.pdf
  • Statistical Analysis Plan (2013-09-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT01985763/SAP_001.pdf